CLINICAL TRIAL: NCT00178763
Title: Phase II Clinical Trial of Cisplatin + Gemcitabine in Combination With Mild, Fever-Range Whole-Body Hyperthermia to Treat Patients With Advanced, Inoperable Pancreatic Cancer
Brief Title: Hyperthermia With Chemotherapy for Locally Advanced or Metastatic Pancreas Cancer
Acronym: FR-WB-TT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Joan M.C Bull, M.D., The University of Texas Health Science Center, Houston
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-02-117
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2011-03-03 (Estimated); Status verified 2011-03

CONDITIONS: Pancreatic Neoplasms
Keywords: Cancer; Pancreatic Cancer; Pancreas; Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms | interventions — Cisplatin; Gemcitabine; Interferon-alpha; peginterferon alfa-2a; Interferon alpha-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): All protocol subjects are treated with fever-range whole-body thermal therapy combined in an optimized schedule with cisplatin + gemcitabine + metronomic low-dose interferon-alpha
  Interventions: Device: Heckel Infrared Radiant Heat Device; Other: cisplatin, gemcitabine, interferon-alpha; Other: thermochemotherapy

INTERVENTIONS:
Device: Heckel Infrared Radiant Heat Device — thermotherapy, maintain a core temperature of 40 degrees centigrade for 6 hours duration
  Other Names: Infrared Radiant Heat Device
Other: cisplatin, gemcitabine, interferon-alpha — cisplatin 60 mg/m2 administered over 3 hours intravenously 36 hours before heat. gemcitabine 600 mg/m2 administered intravenously over 1 hour during 40 degree heat. interferon-alpha 1 million international units subcutaneously daily during protocol.
  Other Names: Cisplatin; Gemzar; Pegasys
Other: thermochemotherapy — fever-range whole-body thermal therapy to 40 degrees centigrade combined with cisplatin 60 mg/m2 + gemcitabine 600 mg/m2 + daily interferon alpha 1 million units.
  Other Names: cisplatin, Cisplatin; gemcitabine, Gemzar; interferon-alpha, Roferon

SUMMARY:
Thermal therapy (hyperthermia, or heat) enhances the chemotherapy anti-tumor kill. Thermal therapy by itself also kills cancer cells. Whole-body thermotherapy is a systemic treatment that includes the entire body. By using fever-range whole-body thermal therapy, cancer cells can be treated wherever they are throughout the entire body. In this study, we are testing a combination of fever-range thermal therapy combined with chemotherapy to test: 1) the response of metastatic or advanced pancreas cancer to the combined modality treatment of thermotherapy and selected chemotherapy; 2) whether it helps the body immunity fight the pancreas cancer; and 3) if this treatment is safe for the patient.

This study does not offer thermal therapy alone. Any patient with measurable, inoperable or metastatic pancreatic cancer may be treated; however, the they will need to undergo specific medical tests to make sure this treatment would be safe for them.

We hypothesize that a combined-modality therapy using fever-range whole-body hyperthermia (FR-WBH; temperature = 40 o C; duration = 6 h), administered in an optimized time/sequence schedule with cisplatin, gemcitabine HCl (gemcitabine), and metronomically administered, low-dose interferon-alpha (IFN-alpha) to patients with inoperable or metastatic pancreas cancer, will, without inducing intolerable toxicity: a.) decrease the pancreatic cancer size; b.) improve quality of life; c.) enhance the immune response against the cancer; d.) increase survival; and e.) allow inoperable pancreatic cancer to be converted to operable disease.

DETAILED DESCRIPTION:
The treatment cycle begins with 6 hours of intravenous (IV) hydration followed by an infusion of the anti-cancer drug, Cisplatin. In addition, at the beginning of this treatment, you will begin low-dose Interferon-alpha injections for the entire duration of your participation in this study. The drug, Interferon-alpha, interrupts the division of cancer cells, destroys tumor blood vessels, and slows tumor growth.

Forty-eight hours after the Cisplatin infusion, you will be treated with fever-range thermal therapy (whole-body hyperthermia, or heat). When your core body temperature reaches 104oF (40oC), a 30-minute (IV) infusion of another chemotherapy drug, gemcitabine (Gemzar) is given. Cisplatin, low-dose Interferon-a and gemcitabine are the only chemotherapy drugs used in this treatment plan. No other chemotherapy drugs are allowed to be given under this treatment plan.

The fever-range whole-body heat treatment is carried out while you are lightly sedated. With this sedation, you will be awake and be able to talk during the treatment, however you will not be uncomfortable. This sedation is used to reduce any discomfort of the 6-hour heat treatment procedure yet will allow you to speak to your nurses.

Your body temperature is raised to 104oF (40oC) over a period of 60-120 minutes. When the body first reaches the target 104oF, we administer the gemcitabine chemotherapy over 60 minutes and continue to maintain the 104 oF body temperature for six hours. At the conclusion of the six hours of thermal treatment, you will be cooled to your normal body temperature, which takes about 30-45 minutes. The entire treatment lasts approximately 8 hours. After the treatment is completed, we will observe you for 2 to 12 hours to make sure you have tolerated the treatment without a problem.

You will continue the low-dose Interferon-alpha. Additionally, you will be given 5-10 days of Leukine (sargramostim) cytokine injections usually beginning 3-5 days after receiving chemotherapy to help support the immune system by helping the body create more white blood cells. White blood cells are important to help your body fight infection.

After treatment, you will need a complete blood count with platelet and differential count each week. These lab studies can be done at your own doctor's office or hospital as long as you make sure that the results are faxed to us. They can also be done in our clinic. We will see you again in approximately three to four weeks and the treatment cycle will be repeated.

We always attempt to perform at least two thermo-chemotherapy cycles. After the second treatment, CT and/or MRI scans are repeated to see if your cancer is smaller. These scans, along with a physical examination and the lab studies, are used to determine if additional heat treatments will be performed. Additional treatments continue based on how well you respond to the treatment. We limit to the number of heat treatments a patient may have using these chemotherapy drugs to a total of six treatments.

ELIGIBILITY:
Inclusion Criteria:

* Candidate must have biopsy-documented locally advanced or metastatic pancreas cancer
* Must be able to successfully complete preliminary function tests
* Must have a good ECOG score
* Must have two functioning lungs

Exclusion Criteria:

* Must not have active metastasis to the brain
* Must not have poor preliminary function tests
* Must not have a low ECOG score
* Must not be taking high-dose corticosteroids
* Must be psychologically stable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2003-09; Primary Completion 2012-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Tumor response, disease-free survival | 2 months to 5 years

SECONDARY OUTCOMES:
Allow inoperable pancreatic cancer to be converted to operable disease | 2 months to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Joan M Bull, M.D., Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Memorial Hermann Hospital, Houston, Texas, United States